CLINICAL TRIAL: NCT00404378
Title: An Open-label, Two Period, Fixed Sequence Study of Healthy Subjects to Assess the Effect of Repeat Oral Dosing of Ketoconazole on the Pharmacokinetics of a Single Oral Dose of [GW679769]
Brief Title: Study Of Healthy Subjects To Assess The Effect Of Ketoconazole And The Way The Body Will React To Casopitant [GW679769]
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKV105093
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: Healthy subjects; Pharmacokinetics; Drug interaction; Ketoconazole; Casopitant
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ketoconazole; casopitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 Treatment Period 1 (Experimental): Subjects will receive single oral dose of 100 milligram (mg) of Casopitant. There will be wash out period of 7 days.
  Interventions: Drug: casopitant 100 mg
- Cohort 1 Treatment Period 2 (Experimental): Subjects will receive ketoconazole 400 mg once daily on Days 1 - 7. On Day 4 subjects will receive a single dose of oral casopitant 100 mg along with ketoconazole.
  Interventions: Drug: ketoconazole; Drug: casopitant 100 mg
- Cohort 2 Treatment Period 1 (Experimental): Subjects will receive single oral dose of 50 mg of Casopitant. There will be wash out period of 7 days.
  Interventions: Drug: Casopitant 50 mg
- Cohort 2 Treatment Period 2 (Experimental): Subjects will receive ketoconazole 400 mg once daily on Days 1 - 7. On Day 4 subjects will receive a single dose of oral casopitant 50 mg along with ketoconazole.
  Interventions: Drug: ketoconazole; Drug: Casopitant 50 mg

INTERVENTIONS:
Drug: ketoconazole — Ketoconazole tablets will be available with dose strength of 200 mg. The dose of ketoconazole 400 mg will be comprised of two 200 mg tablets. On Day 4 of Treatment Period 2, the dose of casopitant and ketoconazole is to be taken at the same time.
  Arms: Cohort 1 Treatment Period 2; Cohort 2 Treatment Period 2
Drug: casopitant 100 mg — Casopitant tablets will be available with dose strength of 50 mg. Subjects will receive two 50 mg tablets for the dose of 100 mg. On Day 4 of Treatment Period 2, the dose of casopitant and ketoconazole is to be taken at the same time
  Other Names: casopitant; ketoconazole
  Arms: Cohort 1 Treatment Period 1; Cohort 1 Treatment Period 2
Drug: Casopitant 50 mg — Casopitant tablets will be available with dose strength of 50 mg and will receive single dose. On Day 4 of Treatment Period 2, the dose of casopitant and ketoconazole is to be taken at the same time.
  Arms: Cohort 2 Treatment Period 1; Cohort 2 Treatment Period 2

SUMMARY:
This is a two period study of healthy adult subjects to characterize the effect of the dosing of ketoconazole on the the way the body reacts to a dose of GW679769, and to assess the safety profile of oral casopitant with and without ketoconazole. This study will consist of a screening period, two treatment periods and a post-treatment follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females
* Females must be of non-childbearing potential
* Adequate organ functions
* Able to swallow and retain oral medications
* Able to understand and comply with study requirements
* Signed ICF

Exclusion Criteria:

* Clinically relevant abnormality identified on the screening exam or any other medical condition or circumstance making the subject unsuitable for participation in the study.
* History of drug or other allergy which contraindicates participation.
* Known immediate hypersensitivity reaction or idiosyncrasy to GW679769 or ketoconazole or drugs chemically related to the study medications.
* Use of an investigational drug within 28 days preceding the first dose of GW679769 or ketoconazole or participation in another clinical trial within the past 30 days.
* Blood donation in excess of 1 pint within 56 days prior to first dose of study medication or intends to donate within 30 days of the post-treatment follow-up visit.
* History of or suspected iron deficiency.
* Positive stool for occult blood.
* Pepsinogen level below the lower limit of laboratory reference range (LLRR).
* Troponin level above 10% of the coefficient of variation of the assay as determined by the laboratory performing the test.
* For male subjects, any history of hypogonadism and treatments associated with hypogonadism including radiation therapy to the testicles.
* For female subjects, a positive serum ß-hCG (beta-human chorionic gonadotropin) pregnancy test.
* Female subject who is lactating.
* Positive urine drug screen (UDS) including alcohol.
* Positive for HIV antibody, hepatitis C antibody or hepatitis B surface antigen
* Positive urinary cotinine. Subjects must not have used any nicotine-containing products, including nicotine patches or gum, within the past 6 months.
* Smoking history = 4 packs per day/year or smoked within the past 12 months.
* History of drug abuse or dependence within the past 6 months.
* History of alcohol abuse within the past 6 months or alcohol consumption in the past 6 months exceeding study requirements
* Presence of uncontrolled nausea & vomiting.
* Presence of an active infection.
* Any degree of heart failure as defined by the New York Heart Association functional classification system.
* Active peptic ulcer disease (PUD) or a history of PUD of unknown etiology.
* Use of any prescription or non-prescription drug(s), herbal or dietary supplements or vitamins within 14 days prior to the first dose of study medication.
* Consumption of any food or drink containing grapefruit or grapefruit juice, apple juice, Seville oranges, kumquats, pomelos or vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi and brussels sprouts, mustard) within 14 days prior to the first dose of study medication.
* History of cholecystectomy or biliary tract disease.
* Any serious or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2006-10-20 (Actual); Primary Completion 2007-01-05 (Actual); Study Completion 2007-01-05 (Actual)

PRIMARY OUTCOMES:
Plasma levels will be measured for casopitant at Period 1: Day 1, 2 & 3. | Period 1: Day 1, 2 & 3
Plasma levels will be measured for casopitant and ketoconazole at Period 2: Day 4, 5, 6, 7, & 8. | Period 2: Day 4, 5, 6, 7, & 8.

SECONDARY OUTCOMES:
clinical lab tests monitoring of International Normalized Ratio (INR) adverse events vital signs 12 lead ECGs liver function tests | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study NKV105093 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/NKV105093?search=study&search_terms=NKV105093#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: NKV105093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKV105093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKV105093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKV105093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKV105093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKV105093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKV105093 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register